CLINICAL TRIAL: NCT00340028
Title: Hormonal Changes in Early Pregnancy: Pilot Study to Evaluate Stored Urine Specimens
Brief Title: Hormonal Changes in Early Pregnancy
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905087; 05-E-N087
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy
Keywords: Ovulation; Diary Record; Urine Collection; Blood Collection; Hormone; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women in Early Pregnancy: Women enrolled in the University of North Carolina's Right from the Start study are followed while trying to become pregnant and through 9 weeks of pregnancy

SUMMARY:
This study will analyze hormones in early pregnancy. Hormonal changes in early pregnancy reflect the quality of implantation in the uterus of the fertilized egg, the function of the corpus luteum (mass of hormone-secreting tissue that forms immediately after ovulation) and placenta, and the health of the embryo. It will determine the following:

* Whether early pregnancy hormones vary by characteristics of the mother
* Whether early pregnancy hormones differ for pregnancies with male or female babies
* Whether early pregnancy hormones can predict the gestational age (age of the baby during pregnancy) and the baby's birth weight
* Hormone activity at the time pregnancy symptoms begin
* How the contribution of the corpus luteum changes during the pregnancy in different women

Stored urine specimens collected from women who participated in the North Carolina Early Pregnancy Study in the 1980s will be used for this study. In addition, to evaluate the quality of the stored samples, new specimens will be collected from women currently enrolled in the University of North Carolina's Right from the Start study. Candidates must be white women not of Latino or Hispanic origin who are between 25 and 35 years of age and who are planning to become pregnant within a few months' time. They must be non-smokers, have regular menstrual cycles, no known fertility problems and no major chronic disease.

Urine specimens are analyzed for hormone levels and other changes in early pregnancy that can be measured in urine. Women providing new urine specimens do the following:

Pre-Pregnancy

The pre-pregnancy part of the study lasts through no more than three consecutive menstrual cycles. Participants who do not become pregnant after three menstrual cycles end the study at that time.

* Have a short interview with a study staff member
* Complete a daily diary, recording any vaginal bleeding or spotting, health status, and use of medications, and mail the diary to the study office once a week
* Use an ovulation testing kit for up to 7 days during their menstrual cycle
* Call the study staff within the first 24 hours of becoming pregnant

Pregnancy

The pregnancy part of the study lasts about 5 weeks.

* Continue to complete daily diary records for weekly pickup by staff member
* Collect urine samples daily and store them in the freezer for weekly pickup by staff member
* Have 1 to 2 tablespoons of blood drawn at home weekly for 4 weeks
* Have a brief follow-up telephone interview around week 12 of their pregnancy

Urine samples are analyzed for hormones such as human chorionic gonadotropin, estrone-3-glucuronide, and pregnanedrol glucuronide. White blood cells are stored for DNA to study such things as genes controlling hormone metabolism.

...

DETAILED DESCRIPTION:
Daily first morning urine specimens were collected throughout the first 8-9 weeks of 151 clinical pregnancies. These specimens are now approximately 20 years in storage, and the stability of markers of placental and corpus luteum function are not known. We will collect new urine specimens for 20 pregnancies to serve as a reference to evaluate the quality of those stored samples.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

We will recruit from the pre-pregnancy participants in the Right From the Start UNC study entitled, Consequences and Course of Uterine Fibroid in Pregnancies.

The women will be selected to be similar to the majority of women in the NC-EPS because we need to have a comparable sample of women in order to best compare hormone levels.

Entry requirements will be:

white (including Hispanic and latino), age 25-35, regular menstrual cycles, nonsmoker (i.e., no smoking in past year), no major chronic disease, no known fertility problems, no more than 3 months of trying for this current pregnancy.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Stored urine specimens collected from women who participated in the North Carolina Early Pregnancy Study in the 1980s will be used for this study. In addition, to evaluate the quality of the stored samples, new specimens will be collected from women currently enrolled in the University of North Carolina's Right from the Start study. Candidates must be white women not of Latino or Hispanic origin who are between 25 and 35 years of age and who are planning to become pregnant within a few months' time. They must be non-smokers, have regular menstrual cycles, no known fertility problems and no major chronic disease.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2005-01-18 (Actual); Primary Completion 2006-02-24 (Actual); Study Completion 2014-04-22 (Actual)

PRIMARY OUTCOMES:
We will assay both old urines and new urines for the estrogen metabolite, the progesterone metabolite, and hCG. | Time points were daily for urine and weekly blood
  no disease treatment monitored

CONTACTS AND LOCATIONS:
Overall Officials: Donna D Baird, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina